CLINICAL TRIAL: NCT01945801
Title: The Effect of Sodium-Restricted Diet and Diuretic in the Severe Sleep Apnea: a Randomized Controlled Trial - DESALT Study
Brief Title: Sodium-Restricted Diet and Diuretic in the Treatment of Severe Sleep Apnea
Acronym: DESALT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GPPG-13-0272; 13-0272 (Other Grant/Funding Number: Fund of Incentive of Research)
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep apnea; Treatment; Sodium-Restricted Diet; Diuretic; Lasilactone
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Spironolactone; Furosemide; Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lasilactone (Active Comparator): Dosage form: One capsule taking in the morning Dosage: furosemide, 20mg, and spironolactone, 100 mg. Frequency and duration: One capsule daily for 7 days.
  Interventions: Drug: Lasilactone
- placebo pill (Placebo Comparator): One capsule taking in the morning. Frequency and duration: One capsule daily for 7 days.
  Interventions: Drug: Placebo
- Sodium-Restricted Diet (Active Comparator): The diet group will receive a regimen with a prescribed intake of three grams of sodium per day
  Interventions: Other: Sodium-Restricted Diet

INTERVENTIONS:
Drug: Lasilactone — Active drug (spironolactone 100 mg plus furosemide 20 mg).
  Other Names: Spironolactone 100 mg plus Furosemide 20 mg
  Arms: Lasilactone
Other: Sodium-Restricted Diet — The sodium-restricted diet will enforce some rules: do not use salt in cooking; do not use the salt shaker; do not ingest any industrialized food; to eat fresh salads and vegetables; do not add high-sodium seasonings, among others. The complete dietary rules will be delivered to each volunteer in a four page handout.
  Other Names: Low sodium diet
  Arms: Sodium-Restricted Diet
Drug: Placebo — The placebo group will receive cellulose-based placebo pills with identical pills and flasks to active drug.
  Other Names: Placebo pill; Control
  Arms: placebo pill

SUMMARY:
This study evaluates the intervention of the 1) sodium-restricted diet, or 2) diuretic, or 3) placebo pill in the treatment of obstructive sleep apnea in adults.

DETAILED DESCRIPTION:
Men with apnea-hypopnea index greater than 30/hour will be included and randomly assigned into three groups: sodium-restricted diet, or diuretic, or control. The intervention will last one week. The diuretic group will receive combined spironolactone 100mg plus furosemide 20mg daily. The diet group will receive a regimen with a maximum intake of three grams of sodium per day. The control group will receive a placebo pill and will maintain all eating habits.

ELIGIBILITY:
Inclusion Criteria:

* Men in the age range from 18 to 60 years
* Full-night in-laboratory polysomnography with apnea-hypopnea index > 30/h in the last three months
* Body mass index < 35 kg/m2
* Informed consent

Exclusion Criteria:

* Already having started any treatment for sleep apnea, including use of continuous positive airway pressure
* NYHA heart failure, any class
* Predominantly central apnea
* Peripheral venous or lymphatic insufficiency
* Any chronic renal disease
* Use of diuretics and substances with action in the central or peripheral nervous system such as benzodiazepines, hypnotics, anticonvulsants, antidepressants, appetite suppressants, amphetamines, antiparkinson agents, muscle relaxants, bronchodilators
* Stroke within 6 months or with incapacitating sequelae
* Any physical, mental or social condition impairing the ability to participate in the trial

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index | One week
  Number of apneas/hour

SECONDARY OUTCOMES:
Somnolence scale (Epworth) and ventilatory parameters | One week
Glycolipid profile | One week
  Total and HDL Cholesterol, Triglycerides, and glucose
Aldosterone Renin Level Activity | One week
  Serum renin and aldosterone
Dosages of urinary 24h | One week
  Aldosterone, sodium, potassium, urea, and creatinine
Inflammatory marker | One week
  C reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Denis Martinez, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre, Universidade Federal do Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Fiori CZ, Martinez D, Montanari CC, Lopez P, Camargo R, Sezera L, Goncalves SC, Fuchs FD. Diuretic or sodium-restricted diet for obstructive sleep apnea-a randomized trial. Sleep. 2018 Apr 1;41(4). doi: 10.1093/sleep/zsy016. PMID 29669139
- [Derived] Fiori CZ, Martinez D, Goncalves SC, Montanari CC, Fuchs FD. Effect of diuretics and sodium-restricted diet on sleep apnea severity: study protocol for a randomized controlled trial. Trials. 2015 Apr 25;16:188. doi: 10.1186/s13063-015-0699-9. PMID 25906818